CLINICAL TRIAL: NCT02479412
Title: A RANDOMIZED, DOUBLE BLIND, MULTIPLE DOSING (14 DAYS), PLACEBO-CONTROLLED, INCOMPLETE BLOCK CROSSOVER, MULTI CENTER STUDY TO ASSESS EFFICACY AND SAFETY OF THREE DOSE LEVELS OF AZD7594, GIVEN ONCE DAILY BY INHALATION, IN PATIENTS WITH MILD TO MODERATE ASTHMA
Brief Title: A Multiple Dosing (14 Days) Study to Assess Efficacy and Safety of Three Dose Levels of AZD7594, Given Once Daily by Inhalation, in Patients With Mild to Moderate Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: D3741C00003; 2014-005306-37 (EudraCT Number)
Record Dates: First submitted 2015-06-17; First posted 2015-06-24 (Estimated); Results first posted 2017-06-23 (Actual); Last update posted 2018-02-15 (Actual); Status verified 2017-08

CONDITIONS: Asthma; Efficacy; Safety
Keywords: Mild to moderate asthma; FEV1; efficacy; safety
MeSH Terms: conditions — Asthma | interventions — velsecorat; Albuterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (9):
- Sequence 1 (Experimental): Placebo once daily for 14 days in Period 1, 58 µg AZD7594 once daily for 14 days in Period 2 and 250 µg AZD7594 once daily for 14 days in Period 3
  Interventions: Drug: 250 µg AZD7594 once daily; Drug: 58 µg AZD7594 once daily; Drug: Placebo once daily; Drug: Salbutamol
- Sequence 2 (Experimental): Placebo once daily for 14 days in Period 1, 250 µg AZD7594 once daily for 14 days in Period 2 and 800 µg AZD7594 once daily for 14 days in Period 3
  Interventions: Drug: 800 μg AZD7594 once daily; Drug: 250 µg AZD7594 once daily; Drug: Placebo once daily; Drug: Salbutamol
- Sequence 3 (Experimental): Placebo once daily for 14 days in Period 1, 800 µg AZD7594 once daily for 14 days in Period 2 and 58 µg AZD7594 once daily for 14 days in Period 3
  Interventions: Drug: 800 μg AZD7594 once daily; Drug: 58 µg AZD7594 once daily; Drug: Placebo once daily; Drug: Salbutamol
- Sequence 4 (Experimental): 58 µg AZD7594 once daily for 14 days in Period 1, Placebo once daily for 14 days in Period 2 and 800 µg AZD7594 once daily for 14 days in Period 3
  Interventions: Drug: 800 μg AZD7594 once daily; Drug: 58 µg AZD7594 once daily; Drug: Placebo once daily; Drug: Salbutamol
- Sequence 6 (Experimental): 250 µg AZD7594 once daily for 14 days in Period 1, Placebo once daily for 14 days in Period 2 and 58 µg AZD7594 once daily for 14 days in Period 3
  Interventions: Drug: 250 µg AZD7594 once daily; Drug: 58 µg AZD7594 once daily; Drug: Placebo once daily; Drug: Salbutamol
- Sequence 8 (Experimental): 800 µg AZD7594 once daily for 14 days in Period 1, Placebo once daily for 14 days in Period 2 and 250 µg AZD7594 once daily for 14 days in Period 3
  Interventions: Drug: 800 μg AZD7594 once daily; Drug: 250 µg AZD7594 once daily; Drug: Placebo once daily; Drug: Salbutamol
- Sequence 5 (Experimental): 58 µg AZD7594 once daily for 14 days in Period 1, 800 µg AZD7594 once daily for 14 days in Period 2 and Placebo once daily for 14 days in Period 3
  Interventions: Drug: 800 μg AZD7594 once daily; Drug: 58 µg AZD7594 once daily; Drug: Placebo once daily; Drug: Salbutamol
- Sequence 7 (Experimental): 250 µg AZD7594 once daily for 14 days in Period 1, 58 µg AZD7594 once daily for 14 days in Period 2 and Placebo once daily for 14 days in Period 3
  Interventions: Drug: 250 µg AZD7594 once daily; Drug: 58 µg AZD7594 once daily; Drug: Placebo once daily; Drug: Salbutamol
- Sequence 9 (Experimental): 800 µg AZD7594 once daily for 14 days in Period 1, 250 µg AZD7594 once daily for 14 days in Period 2 and Placebo once daily for 14 days in Period 3
  Interventions: Drug: 800 μg AZD7594 once daily; Drug: 250 µg AZD7594 once daily; Drug: Placebo once daily; Drug: Salbutamol

INTERVENTIONS:
Drug: 800 μg AZD7594 once daily — Once daily dosing of 800 µg AZD7594 for 14 days; each dose of AZD7594 inhalation powder will be administered via a dry powder monodose inhaler as 2 hard capsules with 2 inhalations per capsule
  Other Names: High dose of AZD7594
  Arms: Sequence 2; Sequence 3; Sequence 4; Sequence 5; Sequence 8; Sequence 9
Drug: 250 µg AZD7594 once daily — Once daily dosing of 800 µg AZD7594 for 14 days; each dose of AZD7594 inhalation powder will be administered via a dry powder monodose inhaler as 2 hard capsules with 2 inhalations per capsule
  Other Names: Medium dose of AZD7594
  Arms: Sequence 1; Sequence 2; Sequence 6; Sequence 7; Sequence 8; Sequence 9
Drug: 58 µg AZD7594 once daily — Once daily dosing of 800 µg AZD7594 for 14 days; each dose of AZD7594 inhalation powder will be administered via a dry powder monodose inhaler as 2 hard capsules with 2 inhalations per capsule
  Other Names: Low dose of AZD7594
  Arms: Sequence 1; Sequence 3; Sequence 4; Sequence 5; Sequence 6; Sequence 7
Drug: Placebo once daily — Once daily dosing of Placebo to AZD7594 for 14 days; each dose of Placebo inhalation powder will be administered via a dry powder monodose inhaler as 2 hard capsules with 2 inhalations per capsule
  Other Names: Placebo
Drug: Salbutamol — Inhalation as needed
  Other Names: Rescue medication

SUMMARY:
This study will be a randomised, double-blind, multiple dose (14 days), placebo-controlled, multi-center study to assess efficacy and safety of three dose levels of AZD7594, given once daily by inhalation, in patients with mild to moderate asthma.

DETAILED DESCRIPTION:
This is a randomized, double-blind, multiple dosing (14 ± 1 days), placebo-controlled, incomplete block crossover, multi-center study to assess efficacy and safety of 3 dose levels of AZD7594, given once daily by inhalation, in patients with mild to moderate asthma.

This multi-center study will be conducted at multiple sites in Europe. It is planned that approximately 48 patients with mild to moderate asthma will be randomized into the study

ELIGIBILITY:
Inclusion Criteria:

* Body mass index of 18 to 35 kg/m2
* Men and women 18 to 75 years of age, inclusive
* Patients need to be non-smokers or ex-smokers (quit ≥ 6 months before the Visit 1) with total smoking history of < 10 pack years
* Documented clinical diagnosis of asthma for ≥ 6 months before the Visit 1
* Patients on low-dose inhaled corticosteroids (ICS) (equivalent of budesonide ≤ 400 μg per day) or low-dose ICS/long-acting β-2 agonist (LABA), or not on any inhaled steroids, or patients on montelukast
* Patients should be controlled on low dose budesonide during the first 14 ±2 days of Run-in Part 1, i.e., they need to have ACQ-5 of ≤ 1.5 at Visit 2.
* Prebronchodilator FEV1 at Visit 3 should be between 40% and 90% of predicted (mean of 2 predose measurements taken 30 minutes apart).
* All patients need to have FeNO concentrations of ≥ 25 parts per billion at Visit 3
* Demonstrate the ability to use the study inhalation device properly
* Women must be of nonchildbearing potential defined as meeting 1 of the following criteria:

  * Permanently or surgically sterilized, including hysterectomy and/or bilateral oophorectomy and/or bilateral salpingectomy
  * Postmenopausal; aged ≤ 50 years and have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and with luteinizing hormone and follicle stimulating hormone levels in the postmenopausal range
  * Postmenopausal; aged > 50 years and have been amenorrheic for 12 months or more, following cessation of all exogenous hormonal treatments
* Male patients should be willing to use a condom to prevent pregnancy and exposure of a female partner to AZD7594 and should refrain from donating sperm or fathering a child from the first day of dosing until 3 months after the last dose of IMP.

Exclusion Criteria:

* Known or suspected hypersensitivity to the IMPs or excipients, including lactose
* Systemic steroid use in the 6 weeks before Visit 1
* Any active disease other than asthma
* Patients on medium to high-dose ICS (equivalent of budesonide > 400 μg per day) or on inhaled anticholinergic combination within the 6 weeks prior to Visit 1
* Compliance with the eDiary of at least 80% of the days is expected in both Run-in and Treatment Periods. Patients with < 80% eDiary compliance during Run-in Periods would not be randomized
* Treatment with biologicals such as monoclonal antibodies or chimeric biomolecules including omalizumab within 6 months or 5 half-lives before Visit 1, whichever is longer
* History or clinical suspicion of any clinically relevant disease or disorder which, in the opinion of the Investigator, may either put the patient at risk because of participation in the study, or influence the results or the patient's ability to participate in the study, or any other safety concerns in the opinion of the Investigator
* ACQ-5 ≥ 3 at any time between Visits 1 and 3
* Any contraindication against the use of vagolytic or sympathomimetic drugs as judged by the Investigator.
* Patients with hepatitis B surface antigen, hepatitis C virus antibody or human immunodeficiency virus (HIV)
* Donation of blood (≥ 450 mL) within 3 months or donation of plasma within 14 days before Visit 1
* Pregnant woman or a nursing mother
* Suspicion of Gilbert's syndrome
* Vulnerable persons (e.g., persons kept in detention)
* ACQ-5 of ≥ 3 or daily rescue use of ≥ 12 puffs for ≥ 3 consecutive days during the enrollment period
* Hypersensitivity to the active substance or to any of the excipients of the Run-in medication (i.e., budesonide)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2015-06-25 (Actual); Primary Completion 2016-02-08 (Actual); Study Completion 2016-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rainard Fuhr, Dr. med., Principal Investigator — PAREXEL International GmbH, Berlin, Germany; Ulrike Westerhausen, Dr., Principal Investigator — Pneumologisches Studienzentrum, Berlin, Germany; Oliver Kornmann, Dr., Principal Investigator — IKF Pneumologie GmbH, Frankfurt, Germany; Jutta Beier, Dr. med., Principal Investigator — Insaf GmbH, Wiesbaden, Germany; Christine Grigat, Dr., Principal Investigator — Clinical Research Hamburg GmbH, Hamburg, Germany; Andrea Ludwig-Sengpiel, Dr., Principal Investigator — KLB Gesundheitsforschung Lübeck GmbH, Lübeck, Germany; Dirk Skowasch, Prof., Principal Investigator — University hospital of Bonn, Department of Internal Medicine II, Bonn, Germany; Anne-Marie Kirsten, Dr., Principal Investigator — Pneumologisches Forschungsinstitut an der LungenClinic Großhansdorf, Großhansdorf, Germany; Tanya Kralimarkova, Dr., Principal Investigator — COMAC Medical Ltd., Sofia, Bulgaria; Anneliese Linnhoff, Dr. med., Principal Investigator — Praxis für Lungen- und Bronchialheilkunde, Allergologie und Umweltmedizin; Margret Jandl, Dr., Principal Investigator — Hamburger Institut für Therapie Forschung GmbH
Locations (7):
- Research Site, Sofia, Bulgaria
- Germany (6):
  - Research Site, Berlin
  - Research Site, Frankfurt
  - Research Site, Großhansdorf
  - Research Site, Hamburg
  - Research Site, Lübeck
  - Research Site, Wiesbaden

REFERENCES:
- [Derived] Brown MN, Fuhr R, Beier J, Su HL, Chen Y, Forsman H, Hamren UW, Jackson H, Aggarwal A. Efficacy and safety of AZD7594, an inhaled non-steroidal selective glucocorticoid receptor modulator, in patients with asthma: a phase 2a randomized, double blind, placebo-controlled crossover trial. Respir Res. 2019 Feb 18;20(1):37. doi: 10.1186/s12931-019-1000-7. PMID 30777086

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in Germany (9 centers) and Bulgaria (1 center). A total of 54 participants with mild to moderate asthma were randomized after screening, and received study treatment (AZD7594 or placebo) given over 3 Treatment Periods in an incomplete block crossover design.
Pre-assignment Details: The study consisted of a 2-part run-in period, 3 treatment periods separated by intervening wash-out periods, and a final period of safety follow-up .
Groups:
- Sequence 1 (Placebo + AZD7594 58 μg + AZD7594 250 μg): Participants received Placebo in Treatment Period 1 (1st intervention - 14 days), AZD7594 58 μg in Treatment Period 2 (2nd intervention - 14 days) and AZD7594 250 μg treatment in Period 3 (3rd intervention - 14 days). After treatment periods 1 and 2, participants had an intervening wash-out period of 21 days.
- Sequence 2 (Placebo + AZD7594 250 μg + AZD7594 800 μg): Participants received Placebo in Treatment Period 1 (1st intervention - 14 days), AZD7594 250 μg in Treatment Period 2 (2nd intervention - 14 days) and AZD7594 800 μg in Treatment Period 3 (3rd intervention - 14 days). After treatment periods 1 and 2, participants had an intervening wash-out period of 21 days.
- Sequence 3 (Placebo + AZD7594 800 µg + AZD7594 58 µg): Participants received Placebo in Treatment Period 1 (1st intervention - 14 days), AZD7594 800 μg in Treatment Period 2 (2nd intervention - 14 days) and AZD7594 58 μg in Treatment Period 3 (3rd intervention - 14 days). After treatment periods 1 and 2, participants had an intervening wash-out period of 21 days.
- Sequence 4 (AZD7594 58 μg + Placebo + AZD7594 800 μg): Participants received AZD7594 58 μg in Treatment Period 1 (1st intervention - 14 days), Placebo in Treatment Period 2 (2nd intervention - 14 days) and AZD7594 800 μg in Treatment Period 3 (3rd intervention - 14 days). After treatment periods 1 and 2, participants had an intervening wash-out period of 21 days.
- Sequence 5 (AZD7594 58 µg + AZD7594 800 µg + Placebo): Participants received AZD7594 58 μg in Treatment Period 1 (1st intervention - 14 days), AZD7594 800 μg in Treatment Period 2 (2nd intervention - 14 days) and Placebo in Treatment Period 3 (3rd intervention - 14 days). After treatment periods 1 and 2, participants had an intervening wash-out period of 21 days.
- Sequence 6 (AZD7594 250 μg + Placebo + AZD7594 58 μg): Participants received AZD7594 250 μg in Treatment Period 1 (1st intervention - 14 days), Placebo in Treatment Period 2 (2nd intervention - 14 days) and AZD7594 58 μg in Treatment Period 3 (3rd intervention - 14 days). After treatment periods 1 and 2, participants had an intervening wash-out period of 21 days.
- Sequence 7 (AZD7594 250 μg + AZD7594 58 μg + Placebo): Participants received AZD7594 250 μg in Treatment Period 1 (1st intervention - 14 days), AZD7594 58 μg in Treatment Period 2 (2nd intervention - 14 days) and Placebo in Treatment Period 3 (3rd intervention- 14 days). After treatment periods 1 and 2, participants had an intervening wash-out period of 21 days.
- Sequence 8 (AZD7594 800 μg + Placebo + AZD7594 250 μg): Participants received AZD7594 800 μg in Treatment Period 1 (1st intervention - 14 days), Placebo in Treatment Period 2 (2nd intervention - 14 days) and AZD7594 250 μg Treatment Period 3 (3rd intervention - 14 days). After treatment periods 1 and 2, participants had an intervening wash-out period of 21 days.
- Sequence 9 (AZD7594 800 μg + AZD7594 250 μg + Placebo): Participant received AZD7594 800 μg in Treatment Period 1 (1st intervention 14 days), AZD7594 250 μg in Treatment Period 2 (2nd intervention - 14 days) and Placebo in Treatment Period 3 (3rd intervention - 14 days). After treatment periods 1 and 2, participants had an intervening wash-out period of 21 days.
Period: Overall Study
Arm/Group | Sequence 1 (Placebo + AZD7594 58 μg + AZD7594 250 μg) | Sequence 2 (Placebo + AZD7594 250 μg + AZD7594 800 μg) | Sequence 3 (Placebo + AZD7594 800 µg + AZD7594 58 µg) | Sequence 4 (AZD7594 58 μg + Placebo + AZD7594 800 μg) | Sequence 5 (AZD7594 58 µg + AZD7594 800 µg + Placebo) | Sequence 6 (AZD7594 250 μg + Placebo + AZD7594 58 μg) | Sequence 7 (AZD7594 250 μg + AZD7594 58 μg + Placebo) | Sequence 8 (AZD7594 800 μg + Placebo + AZD7594 250 μg) | Sequence 9 (AZD7594 800 μg + AZD7594 250 μg + Placebo)
Started | 6 | 6 | 6 | 7 | 6 | 5 | 6 | 5 | 7
Completed | 6 | 6 | 4 | 6 | 5 | 5 | 6 | 4 | 6
Not Completed | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Study-specific withdrawal criteria | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1
Not completed — Randomization to wrong PK sampling group | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1 (Placebo + AZD7594 58 μg + AZD7594 250 μg) | Sequence 2 (Placebo + AZD7594 250 μg + AZD7594 800 μg) | Sequence 3 (Placebo + AZD7594 800 µg + AZD7594 58 µg) | Sequence 4 (AZD7594 58 μg + Placebo + AZD7594 800 μg) | Sequence 5 (AZD7594 58 µg + AZD7594 800 µg + Placebo) | Sequence 6 (AZD7594 250 μg + Placebo + AZD7594 58 μg) | Sequence 7 (AZD7594 250 μg + AZD7594 58 μg + Placebo) | Sequence 8 (AZD7594 800 μg + Placebo + AZD7594 250 μg) | Sequence 9 (AZD7594 800 μg + AZD7594 250 μg + Placebo) | Total
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 6 | 5 | 6 | 5 | 7 | 54
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Age (years) | 49 (14) | 50 (10) | 56 (10) | 50 (17) | 49 (7) | 55 (9) | 48 (14) | 55 (14) | 46 (13) | 51 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 2 | 0 | 3 | 2 | 0 | 1 | 1 | 10
  Male | 5 | 6 | 4 | 7 | 3 | 3 | 6 | 4 | 6 | 44

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of AZD7594 by Assessment of the Change From Baseline in Morning Trough Forced Expiratory Volume in 1 Second (FEV1) on Day 15
Description: Comparison of the efficacy of AZD7594 in terms of change from baseline in morning trough forced expiratory volume in 1 second (FEV1) on Day 15 (defined as the average of the values at 23:00 and 23:30 hours after last dose of investigational medicinal product [IMP] on Day 14) with placebo
Time Frame: On Day 1 (pre-dose) and on Day 15 in each period
Population: All randomized participants who received at least one dose of randomized study drug, were included in the full analysis set (FAS), following the principle of intent to treat (ITT). Participants were included in the analysis according to the treatment to which they were randomized.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Groups:
- AZD7594: AZD7594 DPI once daily
- Placebo: Placebo for AZD7594 DPI once daily
Arm/Group | AZD7594 | Placebo
Number analyzed (Participants) | 33 | 51
Liters
  AZD7594 58 µg vs. PBO | 0.08639 [-0.01650 to 0.1893] | 0.05948 [-0.02453 to 0.1435]
  AZD7594 250 µg vs.PBO | 0.1355 [0.03283 to 0.2382] | 0.05948 [-0.02453 to 0.1435]
  AZD7594 800 µg vs.PBO | 0.2072 [0.1041 to 0.3104] | 0.05948 [-0.02453 to 0.1435]
Statistical Analysis 1: Comparison: AZD7594 vs Placebo; AZD7594 58 µg vs. PBO; Test type: Superiority or Other; p = 0.6379, Mixed Models Analysis; Mean Difference (Final Values) = 0.02691, 95% CI 2-sided [-0.08626 to 0.1401], Standard Error of Mean 0.05697
Statistical Analysis 2: Comparison: AZD7594 vs Placebo; AZD7594 250 µg vs.PBO; Test type: Superiority or Other; p = 0.1827, Mixed Models Analysis; Mean Difference (Final Values) = 0.07604, 95% CI 2-sided [-0.03645 to 0.1885], Standard Error of Mean 0.05663
Statistical Analysis 3: Comparison: AZD7594 vs Placebo; AZD7594 800 μg vs. PBO; Test type: Superiority or Other; p = 0.0108, Mixed Models Analysis; Mean Difference (Final Values) = 0.1478, 95% CI 2-sided [0.03494 to 0.2606], Standard Error of Mean 0.05679

2. Secondary Outcome: Efficacy of AZD7594 by Assessment of the Change From Baseline in Fractional Exhaled Nitric Oxide (FeNO) on Day 8
Description: The efficacy of AZD7594 was assessed in terms of change from baseline in fractional exhaled nitric oxide (FeNO) on Day 8
Time Frame: On Day 1 (pre-dose) and on Day 8 in each period
Population: All randomized participants who received at least one dose of randomized study drug, were included in the FAS, following the principle of ITT. Participants were included in the analysis according to the treatment to which they were randomized.
Measure: Least Squares Mean (95% Confidence Interval); unit: Parts per billion (ppb)
Arm/Group | AZD7594 | Placebo
Number analyzed (Participants) | 33 | 52
Parts per billion (ppb)
  AZD7594 58 (Participant count=32) µg vs. PBO | -9.153 [-15.08 to -3.230] | -4.296 [-9.046 to 0.4536]
  AZD7594 250 µg (Participant count=33) vs. PBO | -14.71 [-20.56 to -8.862] | -4.296 [-9.046 to 0.4536]
  AZD7594 800 µg (Participant count=32) vs. PBO | -19.04 [-24.99 to -13.10] | -4.296 [-9.046 to 0.4536]
Statistical Analysis 1: Comparison: AZD7594 vs Placebo; AZD7594 58 µg vs. PBO; Test type: Superiority or Other; p = 0.1342, Mixed Models Analysis; Mean Difference (Final Values) = -4.857, 95% CI 2-sided [-11.24 to 1.528], Standard Error of Mean 3.214
Statistical Analysis 2: Comparison: AZD7594 vs Placebo; AZD7594 250 µg vs. PBO; Test type: Superiority or Other; p = 0.0016, Mixed Models Analysis; Mean Difference (Final Values) = -10.41, 95% CI 2-sided [-16.75 to -4.075], Standard Error of Mean 3.190
Statistical Analysis 3: Comparison: AZD7594 vs Placebo; AZD7594 800 µg vs. PBO; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -14.75, 95% CI 2-sided [-21.18 to -8.319], Standard Error of Mean 3.236

3. Secondary Outcome: Efficacy of AZD7594 by Assessment of the Change From Baseline in Fractional Exhaled Nitric Oxide (FeNO) on Day 15
Description: The efficacy of AZD7594 was assessed in terms of change from baseline in fractional exhaled nitric oxide (FeNO) on Day 15
Time Frame: On Day 1 (pre-dose) and on Day 15 in each period
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Parts per billion (ppb)
Arm/Group | AZD7594 | Placebo
Number analyzed (Participants) | 33 | 51
Parts per billion (ppb)
  AZD7594 58 µg (Participant count=32) vs. PBO | -14.40 [-22.67 to -6.129] | -0.5488 [-6.723 to 5.626]
  AZD7594 250 µg (Participant count=33) vs. PBO | -14.81 [-22.96 to -6.657] | -0.5488 [-6.723 to 5.626]
  AZD7594 800 µg (Participant count=32) vs. PBO | -20.44 [-28.72 to -12.17] | -0.5488 [-6.723 to 5.626]
Statistical Analysis 1: Comparison: AZD7594 vs Placebo; AZD7594 58 µg vs. PBO; Test type: Superiority or Other; p = 0.0084, Mixed Models Analysis; Mean Difference (Final Values) = -13.85, 95% CI 2-sided [-24.06 to -3.642], Standard Error of Mean 5.139
Statistical Analysis 2: Comparison: AZD7594 vs Placebo; AZD7594 250 µg vs. PBO; Test type: Superiority or Other; p = 0.0062, Mixed Models Analysis; Mean Difference (Final Values) = -14.26, 95% CI 2-sided [-24.37 to -4.149], Standard Error of Mean 5.088
Statistical Analysis 3: Comparison: AZD7594 vs Placebo; AZD7594 800 µg vs. PBO; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; Mean Difference (Final Values) = -19.90, 95% CI 2-sided [-30.10 to -9.689], Standard Error of Mean 5.137

4. Secondary Outcome: Efficacy of AZD7594 by Assessment of the Change From Baseline in Trough Forced Expiratory Volume in 1 Second (FEV1) on Day 8
Description: The efficacy of AZD7594 was assessed in terms of change from baseline in morning trough forced expiratory volume in 1 second (FEV1) on Day 8 (defined as the average of the values at 23:00 and 23:30 hours after last dose of investigational medicinal product [IMP] on Day 7)
Time Frame: On Day 1 (pre-dose) and on Day 8 (pre-dose) in each period
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | AZD7594 | Placebo
Number analyzed (Participants) | 33 | 52
Liters
  AZD7594 58 μg vs. PBO | 0.1016 [-0.00007235 to 0.2033] | 0.07112 [-0.009222 to 0.1515]
  AZD7594 250 μg vs. PBO | 0.08856 [-0.01295 to 0.1901] | 0.07112 [-0.009222 to 0.1515]
  AZD7594 800 μg vs. PBO | 0.2272 [0.1252 to 0.3293] | 0.07112 [-0.009222 to 0.1515]
Statistical Analysis 1: Comparison: AZD7594 vs Placebo; AZD7594 58 μg vs. PBO; Test type: Superiority or Other; p = 0.6036, Mixed Models Analysis; Mean Difference (Final Values) = 0.03051, 95% CI 2-sided [-0.08579 to 0.1468], Standard Error of Mean 0.05856
Statistical Analysis 2: Comparison: AZD7594 vs Placebo; AZD7594 250 μg vs. PBO; Test type: Superiority or Other; p = 0.7670, Mixed Models Analysis; Mean Difference (Final Values) = 0.01744, 95% CI 2-sided [-0.09912 to 0.1340], Standard Error of Mean 0.05869
Statistical Analysis 3: Comparison: AZD7594 vs Placebo; AZD7594 800 μg vs. PBO; Test type: Superiority or Other; p = 0.0093, Mixed Models Analysis; Mean Difference (Final Values) = 0.1561, 95% CI 2-sided [0.03943 to 0.2728], Standard Error of Mean 0.05874

5. Secondary Outcome: Efficacy of AZD7594 by Assessment of the Change From Baseline in Trough Forced Vital Capacity (FVC) on Day 15
Description: The efficacy of AZD7594 was assessed in terms of change from baseline in morning trough forced vital capacity (FVC) on Day 15 (defined as the average of the values at 23:00 and 23:30 hours after last dose of investigational medicinal product [IMP] on Day 14)
Time Frame: On Day 1 (pre-dose) and on Day 15 (pre-dose) in each period
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | AZD7594 | Placebo
Number analyzed (Participants) | 33 | 51
Liters
  AZD7594 58 μg vs. PBO | 0.04186 [-0.06673 to 0.1505] | 0.07653 [-0.01626 to 0.1693]
  AZD7594 250 μg vs. PBO | 0.1047 [-0.003607 to 0.2131] | 0.07653 [-0.01626 to 0.1693]
  AZD7594 800 μg vs. PBO | 0.1382 [0.02938 to 0.2471] | 0.0765 [-0.01626 to 0.1693]
Statistical Analysis 1: Comparison: AZD7594 vs Placebo; AZD7594 58 μg vs. PBO; Test type: Superiority or Other; p = 0.5207, Mixed Models Analysis; Mean Difference (Final Values) = -0.03467, 95% CI 2-sided [-0.1415 to 0.07213], Standard Error of Mean 0.05377
Statistical Analysis 2: Comparison: AZD7594 vs Placebo; AZD7594 250 μg vs. PBO; Test type: Superiority or Other; p = 0.5983, Mixed Models Analysis; Mean Difference (Final Values) = 0.02821, 95% CI 2-sided [-0.07778 to 0.1342], Standard Error of Mean 0.05336
Statistical Analysis 3: Comparison: AZD7594; AZD7594 800 μg vs. PBO; Test type: Superiority or Other; p = 0.2538, Mixed Models Analysis; Mean Difference (Final Values) = 0.06169, 95% CI 2-sided [-0.04501 to 0.1684], Standard Error of Mean 0.05371

6. Secondary Outcome: Efficacy of AZD7594 by Assessment of the Change From Baseline in Trough Forced Vital Capacity (FVC) on Day 8
Description: The efficacy of AZD7594 was assessed in terms of change from baseline in morning trough forced vital capacity (FVC) on Day 8 (defined as the average of the values at 23:00 and 23:30 hours after last dose of investigational medicinal product [IMP] on Day 7)
Time Frame: On Day 1 (pre-dose) and on Day 8 (pre-dose) in each period
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | AZD7594 | Placebo
Number analyzed (Participants) | 33 | 52
Liters
  AZD7594 58 μg vs. PBO | 0.06179 [-0.04132 to 0.1649] | 0.08441 [0.001635 to 0.1672]
  AZD7594 250 μg vs. PBO | 0.08410 [-0.01877 to 0.1870] | 0.08441 [0.001635 to 0.1672]
  AZD7594 800 μg vs. PBO | 0.1527 [0.04929 to 0.2562] | 0.08441 [0.001635 to 0.1672]
Statistical Analysis 1: Comparison: AZD7594 vs Placebo; AZD7594 58 μg vs. PBO; Test type: Superiority or Other; p = 0.6945, Mixed Models Analysis; Mean Difference (Final Values) = -0.02262, 95% CI 2-sided [-0.1367 to 0.09144], Standard Error of Mean 0.05743
Statistical Analysis 2: Comparison: AZD7594 vs Placebo; AZD7594 250 μg vs. PBO; Test type: Superiority or Other; p = 0.9957, Mixed Models Analysis; Mean Difference (Final Values) = -0.000314, 95% CI 2-sided [-0.1146 to 0.1140], Standard Error of Mean 0.05755
Statistical Analysis 3: Comparison: AZD7594 vs Placebo; AZD7594 800 μg vs. PBO; Test type: Superiority or Other; p = 0.2398, Mixed Models Analysis; Mean Difference (Final Values) = 0.06831, 95% CI 2-sided [-0.04637 to 0.1830], Standard Error of Mean 0.05774

7. Secondary Outcome: Efficacy of AZD7594 by Assessment of the Change From Baseline in Morning Peak Expiratory Flow (mPEF) Before Administration Over the Treatment Period
Description: The efficacy of AZD7594 was assessed in terms of change from baseline in morning peak expiratory flow (mPEF) before administration of the investigational medicinal product (IMP) in each treatment period. The first PEF measurement was on the evening of Visit 1. Every morning and every evening after Visit 1, patients were required to perform 3 maneuvers for PEF assessment. The highest value from among the 3 assessments was marked as mPEF with the date and time of the measurement. The final PEF assessment was done on the morning of Visit 11 (Day 15 of Treatment Period 3).
Time Frame: Every morning at pre-dose from Day 1 to Day 15
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: L/min
Arm/Group | AZD7594 | Placebo
Number analyzed (Participants) | 33 | 52
L/min
  AZD7594 58 μg vs. PBO | 10.42 [-1.909 to 22.74] | 0.08136 [-10.50 to 10.66]
  AZD7594 250 μg vs. PBO | 5.334 [-6.975 to 17.64] | 0.08136 [-10.50 to 10.66]
  AZD7594 800 μg vs. PBO | 12.60 [0.2402 to 24.96] | 0.08136 [-10.50 to 10.66]
Statistical Analysis 1: Comparison: AZD7594 vs Placebo; AZD7594 58 μg vs. PBO; Test type: Superiority or Other; p = 0.0819, Mixed Models Analysis; Mean Difference (Final Values) = 10.34, 95% CI 2-sided [-1.335 to 22.01], Standard Error of Mean 5.877
Statistical Analysis 2: Comparison: AZD7594 vs Placebo; AZD7594 250 μg vs. PBO; Test type: Superiority or Other; p = 0.3741, Mixed Models Analysis; Mean Difference (Final Values) = 5.253, 95% CI 2-sided [-6.427 to 16.93], Standard Error of Mean 5.881
Statistical Analysis 3: Comparison: AZD7594 vs Placebo; AZD7594 800 μg vs. PBO; Test type: Superiority or Other; p = 0.0374, Mixed Models Analysis; Mean Difference (Final Values) = 12.52, 95% CI 2-sided [0.7481 to 24.29], Standard Error of Mean 5.926

8. Secondary Outcome: Efficacy of AZD7594 by Assessment of the Change From Baseline in Evening Peak Expiratory Flow (ePEF) Before Administration Over the Treatment Period
Description: The efficacy of AZD7594 was assessed in terms of change from baseline in evening peak expiratory flow (ePEF) in each treatment period. The first PEF measurement was on the evening of Visit 1. Every morning and every evening after Visit 1, patients were required to perform 3 maneuvers for PEF assessment. The highest value from among the 3 assessments was marked as ePEF together with the date and time of the measurement. The final PEF assessment was done on the morning of Visit 11 (Day 15 of Treatment Period 3).
Time Frame: Every evening from Day 1 to Day 14 in each period
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: L/min
Arm/Group | AZD7594 | Placebo
Number analyzed (Participants) | 33 | 51
L/min
  AZD7594 58 μg vs. PBO | 7.475 [-4.426 to 19.38] | -8.257 [-18.71 to 2.193]
  AZD7594 250 μg vs. PBO | 6.040 [-5.839 to 17.92] | -8.257 [-18.71 to 2.193]
  AZD7594 800 μg vs. PBO | 11.65 [-0.2692 to 23.58] | -8.257 [-18.71 to 2.193]
Statistical Analysis 1: Comparison: AZD7594 vs Placebo; AZD7594 58 μg vs. PBO; Test type: Superiority or Other; p = 0.0044, Mixed Models Analysis; Mean Difference (Final Values) = 15.73, 95% CI 2-sided [5.039 to 26.43], Standard Error of Mean 5.384
Statistical Analysis 2: Comparison: AZD7594 vs Placebo; AZD7594 250 μg vs. PBO; Test type: Superiority or Other; p = 0.0098, Mixed Models Analysis; Mean Difference (Final Values) = 14.30, 95% CI 2-sided [3.534 to 25.06], Standard Error of Mean 5.419
Statistical Analysis 3: Comparison: AZD7594 vs Placebo; AZD7594 800 μg vs. PBO; Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis; Mean Difference (Final Values) = 19.91, 95% CI 2-sided [9.068 to 30.75], Standard Error of Mean 5.459

9. Secondary Outcome: Efficacy of AZD7594 by Assessment of the Change From Baseline in Average Daily Use of Rescue Salbutamol Over the Treatment Period
Description: The efficacy of AZD7594 was assessed in terms of change from baseline in average daily use of salbutamol (each morning and evening) in each treatment period.
Time Frame: Every day from Day 1 to Day 15 (from evening of Day 1 to morning of Day 15)
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Number of inhalations per day
Arm/Group | AZD7594 | Placebo
Number analyzed (Participants) | 33 | 51
Number of inhalations per day
  AZD7594 58 μg vs. PBO | -0.6776 [-1.071 to -0.2841] | -0.3340 [-0.6733 to 0.005227]
  AZD7594 250 μg vs. PBO | -0.8193 [-1.212 to -0.4267] | -0.3340 [-0.6733 to 0.005227]
  AZD7594 800 μg vs. PBO | -1.137 [-1.531 to -0.7422] | -0.3340 [-0.6733 to 0.005227]
Statistical Analysis 1: Comparison: AZD7594 vs Placebo; AZD7594 58 μg vs. PBO; Test type: Superiority or Other; p = 0.0723, Mixed Models Analysis; Mean Difference (Final Values) = -0.3435, 95% CI 2-sided [-0.7189 to 0.03179], Standard Error of Mean 0.1890
Statistical Analysis 2: Comparison: AZD7594 vs Placebo; AZD7594 250 μg vs. PBO; Test type: Superiority or Other; p = 0.0124, Mixed Models Analysis; Mean Difference (Final Values) = -0.4852, 95% CI 2-sided [-0.8631 to -0.1073], Standard Error of Mean 0.1903
Statistical Analysis 3: Comparison: AZD7594 vs Placebo; AZD7594 800 μg vs. PBO; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -0.8026, 95% CI 2-sided [-1.183 to -0.4224], Standard Error of Mean 0.1914

10. Secondary Outcome: Efficacy of AZD7594 by Assessment of the Change From Baseline to Day 15 in Asthma Control Questionnaire-5
Description: The efficacy of AZD7594 was assessed in terms of change from baseline to Day 15 in Asthma Control Questionnaire-5 in each treatment period. Five questions were asked and each question was scored on a scale of 0 to 6, where a higher score represents a more severe impairment/symptom. The ACQ-5 score at a given visit was defined as the average of the scores given for each of the questions, calculated as ACQ-5 score = Sum of 5 scores/5.
Time Frame: At baseline and on Day 15 in each period
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Unit on a scale
Arm/Group | AZD7594 | Placebo
Number analyzed (Participants) | 33 | 52
Unit on a scale
  AZD7594 58 μg vs. PBO | -0.2929 [-0.4744 to -0.1113] | 0.01428 [-0.1281 to 0.1567]
  AZD7594 250 μg vs. PBO | -0.1681 [-0.3496 to 0.01335] | 0.1428 [-0.1281 to 0.1567]
  AZD7594 800 μg vs. PBO | -0.4158 [-0.5975 to -0.2342] | 0.01428 [-0.1281 to 0.1567]
Statistical Analysis 1: Comparison: AZD7594 vs Placebo; AZD7594 58 μg vs. PBO; Test type: Superiority or Other; p = 0.0044, Mixed Models Analysis; Mean Difference (Final Values) = -0.3071, 95% CI 2-sided [-0.5159 to -0.09836], Standard Error of Mean 0.1051
Statistical Analysis 2: Comparison: AZD7594 vs Placebo; AZD7594 250 μg vs. PBO; Test type: Superiority or Other; p = 0.0883, Mixed Models Analysis; Mean Difference (Final Values) = -0.1824, 95% CI 2-sided [-0.3927 to 0.02789], Standard Error of Mean 0.1059
Statistical Analysis 3: Comparison: AZD7594 vs Placebo; AZD7594 800 μg vs. PBO; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -0.4301, 95% CI 2-sided [-0.6397 to -0.2205], Standard Error of Mean 0.1055

11. Secondary Outcome: Efficacy of AZD7594 by Assessment of the Change From Baseline to Day 8 in Asthma Control Questionnaire-5
Description: The efficacy of AZD7594 was assessed in terms of change from baseline to Day 15 in Asthma Control Questionnaire-5 in each treatment period. Five questions were asked and each question was scored on a scale of 0 to 6, where a lower score represents a more severe impairment/symptom. The ACQ-5 score at a given visit was defined as the average of the scores given for each of the questions, calculated as ACQ-5 score = Sum of 5 scores/5.
Time Frame: At baseline and on Day 8 in each period
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Unit on a scale
Arm/Group | AZD7594 | Placebo
Number analyzed (Participants) | 33 | 52
Unit on a scale
  AZD7594 58 μg vs. PBO | -0.2724 [-0.4309 to -0.1138] | -0.1072 [-0.2320 to 0.01748]
  AZD7594 250 μg vs. PBO | -0.1980 [-0.3565 to -0.03952] | -0.1072 [-0.2320 to 0.01748]
  AZD7594 800 μg vs. PBO | -0.3604 [-0.5191 to -0.2017] | -0.1072 [-0.2320 to 0.01748]
Statistical Analysis 1: Comparison: AZD7594 vs Placebo; AZD7594 58 μg vs. PBO; Test type: Superiority or Other; p = 0.0741, Mixed Models Analysis; Mean Difference (Final Values) = -0.1651, 95% CI 2-sided [-0.3466 to 0.01638], Standard Error of Mean 0.09139
Statistical Analysis 2: Comparison: AZD7594 vs Placebo; AZD7594 250 μg vs. PBO; Test type: Superiority or Other; p = 0.3265, Mixed Models Analysis; Mean Difference (Final Values) = -0.09079, 95% CI 2-sided [-0.2736 to 0.09201], Standard Error of Mean 0.09204
Statistical Analysis 3: Comparison: AZD7594 vs Placebo; AZD7594 800 μg vs. PBO; Test type: Superiority or Other; p = 0.0070, Mixed Models Analysis; Mean Difference (Final Values) = -0.2532, 95% CI 2-sided [-0.4354 to -0.07092], Standard Error of Mean 0.09176

12. Secondary Outcome: Efficacy of AZD7594 by Assessment of Night-time Awakenings
Description: The efficacy of AZD7594 was assessed in terms of change in nighttime awakenings in each treatment period. The patients were asked to answer 'Yes' or 'No' to the question of "Did your asthma cause you to wake up last night?". If yes, the number and percentage of days that had a night-time awakening were determined for each of the study periods.
Time Frame: At baseline and from Day 2 to Day 15 in each period
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Number of nighttime awakenings
Arm/Group | AZD7594 | Placebo
Number analyzed (Participants) | 33 | 52
Number of nighttime awakenings
  AZD7594 58 μg vs. PBO | -0.4120 [-0.7229 to -0.1010] | 0.006541 [-0.2509 to 0.2640]
  AZD7594 250 μg vs. PBO | -0.1729 [-0.4833 to 0.1376] | 0.006541 [-0.2509 to 0.2640]
  AZD7594 800 μg vs. PBO | -0.7595 [-1.071 to -0.4479] | 0.006541 [-0.2509 to 0.2640]
Statistical Analysis 1: Comparison: AZD7594 vs Placebo; AZD7594 58 μg vs. PBO; Test type: Superiority or Other; p = 0.0116, Mixed Models Analysis; Mean Difference (Final Values) = -0.4185, 95% CI 2-sided [-0.7414 to -0.09563], Standard Error of Mean 0.1626
Statistical Analysis 2: Comparison: AZD7594 vs Placebo; AZD7594 250 μg vs. PBO; Test type: Superiority or Other; p = 0.2732, Mixed Models Analysis; Mean Difference (Final Values) = -0.1794, 95% CI 2-sided [-0.5027 to 0.1438], Standard Error of Mean 0.1628
Statistical Analysis 3: Comparison: AZD7594 vs Placebo; AZD7594 800 μg vs. PBO; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -0.7661, 95% CI 2-sided [-1.091 to -0.4411], Standard Error of Mean 0.1636

13. Secondary Outcome: Efficacy of AZD7594 by Assessment of Daily Symptom Score
Description: The efficacy of AZD7594 was assessed in terms of change in daily symptom score from baseline to average of treatment period post dose (Day 1-14) in each treatment period. Severity scores for asthma symptoms were recorded twice daily, once in the morning and once in the evening with the scoring system of 0-no asthma symptoms, 1-toleratable asthma symptoms, 2-discomfort asthma symptoms with normal activities (or with sleep) and 3-asthma symptoms with impaired normal activities (or to sleep).
Time Frame: At baseline and from Day 1 to Day 14 in each period
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Unit on a scale
Arm/Group | AZD7594 | Placebo
Number analyzed (Participants) | 33 | 51
Unit on a scale
  AZD7594 58 μg vs. PBO | -0.1190 [-0.2190 to -0.01903] | -0.01229 [-0.09729 to 0.07270]
  AZD7594 250 μg vs. PBO | -0.09435 [-0.1941 to 0.005411] | -0.01229 [-0.09729 to 0.07270]
  AZD7594 800 μg vs. PBO | -0.2150 [-0.3151 to -0.1149] | -0.01229 [-0.09729 to 0.07270]
Statistical Analysis 1: Comparison: AZD7594 vs Placebo; AZD7594 58 μg vs. PBO; Test type: Superiority or Other; p = 0.0349, Mixed Models Analysis; Mean Difference (Final Values) = -0.1067, 95% CI 2-sided [-0.2057 to -0.007755], Standard Error of Mean 0.04982
Statistical Analysis 2: Comparison: AZD7594 vs Placebo; AZD7594 250 μg vs. PBO; Test type: Superiority or Other; p = 0.1052, Mixed Models Analysis; Mean Difference (Final Values) = -0.08205, 95% CI 2-sided [-0.1817 to 0.01756], Standard Error of Mean 0.05015
Statistical Analysis 3: Comparison: AZD7594 vs Placebo; AZD7594 800 μg vs. PBO; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -0.2027, 95% CI 2-sided [-0.3028 to -0.1025], Standard Error of Mean 0.05044

14. Secondary Outcome: Efficacy of AZD7594 by Assessment of Asthma Control Days
Description: The efficacy of AZD7594 was assessed in terms of amount of asthma control days in each treatment period. An asthma control day was defined as a day with asthma symptom score = 0, a night with no awakenings due to asthma symptoms and a day with no use of rescue medication. A given calendar day was defined as an asthma control day if it fulfills the criteria for a symptom-free day and for a rescue medication-free day
Time Frame: At baseline and from Day 1 to Day 14 post-dose in each period
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Asthma control days
Arm/Group | AZD7594 | Placebo
Number analyzed (Participants) | 33 | 51
Asthma control days
  AZD7594 58 μg vs. PBO | 0.9502 [0.3166 to 1.584] | 0.2773 [-0.2745 to 0.8290]
  AZD7594 250 μg vs. PBO | 0.705 [0.07299 to 1.338] | 0.2773 [-0.2745 to 0.8290]
  AZD7594 800 μg vs. PBO | 1.219 [0.5843 to 1.853] | 0.2773 [-0.2745 to 0.8290]
Statistical Analysis 1: Comparison: AZD7594 vs Placebo; AZD7594 58 μg vs. PBO; Test type: Superiority or Other; p = 0.0247, Mixed Models Analysis; Mean Difference (Final Values) = 0.6730, 95% CI 2-sided [0.08779 to 1.258], Standard Error of Mean 0.2946
Statistical Analysis 2: Comparison: AZD7594 vs Placebo; AZD7594 250 μg vs. PBO; Test type: Superiority or Other; p = 0.1521, Mixed Models Analysis; Mean Difference (Final Values) = 0.4281, 95% CI 2-sided [-0.1607 to 1.017], Standard Error of Mean 0.2965
Statistical Analysis 3: Comparison: AZD7594 vs Placebo; AZD7594 800 μg vs. PBO; Test type: Superiority or Other; p = 0.0022, Mixed Models Analysis; Mean Difference (Final Values) = 0.9415, 95% CI 2-sided [0.3483 to 1.535], Standard Error of Mean 0.2987

15. Secondary Outcome: Number of Participants With Adverse Events
Description: Assessment of safety and tolerability of three dose levels of AZD7594 in participants with mild to moderate asthma. IP referred to investigational product.
Time Frame: From Screening to Follow-up (these two examinations are up to 165 days apart)
Population: The safety analysis set (SAF) included all randomized participants who received at least one dose of randomized study drug during the treatment periods of the study. This analysis set was classified by actual treatment received. If no participants received incorrect treatment then the SAF was identical to the FAS.
Measure: Number; unit: Number of participants
Groups:
- AZD7594 58 μg: AZD7594 DPI once daily - 2 capsules of 29 μg
- AZD7594 250 μg: AZD7594 DPI once daily - 2 capsules of 125 μg
- AZD7594 800 μg: AZD7594 DPI once daily - 2 capsules of 400 μg
Arm/Group | Placebo | AZD7594 58 μg | AZD7594 250 μg | AZD7594 800 μg
Number analyzed (Participants) | 52 | 34 | 34 | 34
Number of participants
  Any AE | 17 | 13 | 9 | 12
  AE causally related to IP | 3 | 1 | 1 | 2
  Any AE with an outcome of death | 0 | 0 | 0 | 0
  Any SAE (including events with outcome of death) | 0 | 0 | 0 | 0
  Any AE leading to discontinuation of IP | 1 | 0 | 0 | 0

16. Secondary Outcome: Rate and Extent of Absorption of Three Dose Levels of AZD7594 by Assessment of Cmax of AZD7594
Description: Comparison of Cmax (maximum observed plasma concentration) of AZD7594 on Day 1 of each treatment period; up to 6 samples were collected in each period (i.e. in participants with intensive pharmacokinetic assessments, at pre-dose and 15 and 30 minutes, and 1, 2, and 4 h post-dose)
Time Frame: On Day 1 in each period (in participants with intensive pharmacokinetic assessments, at pre-dose and 15 and 30 minutes, and 1, 2, and 4 h post-dose)
Population: The PK analysis set (PKS) included the subset of all randomized participants for whom 24-hour PK sampling was performed on Day 14, for whom the primary PK parameters (Cmax , AUC(0-4), Cmax,ss, AUC(0-24)) were calculated in at least one treatment period, and who had no major protocol deviations considered to impact the analysis of the PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol/L
Arm/Group | AZD7594 58 μg | AZD7594 250 μg | AZD7594 800 μg
Number analyzed (Participants) | 9 | 9 | 8
pmol/L | 36.40 (32.80) | 92.02 (34.17) | 169.7 (43.21)

17. Secondary Outcome: Rate and Extent of Absorption of Three Dose Levels of AZD7594 by Assessment of AUC(0-4) of AZD7594
Description: Comparison of AUC(0-4) (Area under the plasma concentration-time curve from time zero to 4 hours after administration) of AZD7594 on Day 1 of each treatment period; up to 6 samples were collected in each period (i.e. in participants with intensive pharmacokinetic assessments, at pre-dose and 15 and 30 minutes, and 1, 2, and 4 h post-dose).
Time Frame: as for outcome 16
Population: The subset of all randomized participants; 24-hour PK sampling was performed on Day 14, the primary PK parameters (Cmax , AUC(0-4), Cmax,ss, AUC(0-24)) were calculated in at least one treatment period, and who had no major protocol deviations considered to impact the analysis of the PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pmol/L
Arm/Group | AZD7594 58 μg | AZD7594 250 μg | AZD7594 800 μg
Number analyzed (Participants) | 9 | 9 | 8
h*pmol/L | 85.02 (8.21) | 188.4 (30.58) | 371.1 (31.55)

18. Secondary Outcome: Rate and Extent of Absorption of Three Dose Levels of AZD7594 Following Multiple Dose Administration by Assessment of Cmax,ss of AZD7594
Description: Comparison of Cmax,ss (observed maximum plasma concentration at steady state) of AZD7594 on Day 14 of each treatment period; up to 10 samples were collected in each period (i.e. in participants with intensive pharmacokinetic assessments, at pre-dose and 15 and 30 minutes, and 1, 2, 4, 8, 12, 16 and 24 h post-dose)
Time Frame: On Day 14 in each period (in participants with intensive pharmacokinetic assessments, at pre-dose and 15 and 30 minutes, and 1, 2, 4, 8, 12, 16 and 24 h post-dose)
Population: PKS included the subset of all randomized participants for whom 24-hour PK sampling was performed on Day 14, for whom the primary PK parameters (Cmax , AUC(0-4), Cmax,ss, AUC(0-24)) were calculated in at least one treatment period, and who had no major protocol deviations considered to impact the analysis of the PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol/L
Arm/Group | AZD7594 58 μg | AZD7594 250 μg | AZD7594 800 μg
Number analyzed (Participants) | 9 | 9 | 8
pmol/L | 54.97 (19.70) | 158.7 (35.01) | 421.6 (37.26)
Statistical Analysis 1: Comparison: AZD7594 58 μg; AZD7594 250 μg versus AZD7594 58 μg; Test type: Superiority or Other; p < 0.0001, ANOVA; Ratio Estimate (%) = 272.20, 90% CI 2-sided [237.43 to 312.05]
Statistical Analysis 2: Comparison: AZD7594 58 μg; AZD7594 800 μg versus AZD7594 58 μg; Test type: Superiority or Other; p < 0.0001, ANOVA; Ratio Estimate (%) = 676.13, 90% CI 2-sided [580.91 to 786.95]

19. Secondary Outcome: Rate and Extent of Absorption of Three Dose Levels of AZD7594 Following Multiple Dose Administration by Assessment of AUC(0-24) of AZD7594
Description: Comparison of AUC(0-24) (Area under the plasma concentration-time curve from time zero to 24 hours after administration) of AZD7594 on Day 14 of each treatment period; up to 10 samples were collected in each period (i.e. in participants with intensive pharmacokinetic assessments, at pre-dose and 15 and 30 minutes, and 1, 2, 4, 8, 12, 16 and 24 h post-dose)
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pmol/L
Arm/Group | AZD7594 58 μg | AZD7594 250 μg | AZD7594 800 μg
Number analyzed (Participants) | 9 | 9 | 8
h*pmol/L | 467.1 (17.91) | 1725 (44.33) | 4894 (52.48)
Statistical Analysis 1: Comparison: AZD7594 58 μg; AZD7594 250 μg versus AZD7594 58 μg; Test type: Superiority or Other; p < 0.0001, ANOVA; Ratio Estimate (%) = 337.82, 90% CI 2-sided [290.80 to 392.43]
Statistical Analysis 2: Comparison: AZD7594 58 μg; AZD7594 800 μg versus AZD7594 58 μg; Test type: Superiority or Other; p < 0.0001, ANOVA; Ratio Estimate (%) = 964.62, 90% CI 2-sided [816.13 to 1140.13]

20. Secondary Outcome: Rate and Extent of Absorption of Three Dose Levels of AZD7594 Following Multiple Dose Administration by Assessment of AUC(0-last) of AZD7594
Description: Comparison of AUC(0-last) (Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration (Day 1 and Day 14)) of AZD7594 (i.e. in participants with intensive pharmacokinetic assessments)
Time Frame: On Day 1 and Day 14 in each period (in participants with intensive pharmacokinetic assessments, on Day 1 at pre-dose and 15 and 30 minutes, and 1, 2 and 4 h post-dose, on Day 14 at pre-dose and 15 and 30 minutes, and 1, 2, 4, 8, 12, 16 and 24 h post-dose)
Population: as for outcome 18
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pmol/L
Arm/Group | AZD7594 58 μg | AZD7594 250 μg | AZD7594 800 μg
Number analyzed (Participants) | 9 | 9 | 8
h*pmol/L
  Day 1 | 56.85 (45.40) | 188.5 (30.57) | 371.8 (31.63)
  Day 14 | 467.3 (17.93) | 1728 (44.36) | 4897 (52.48)

21. Secondary Outcome: Rate and Extent of Absorption of Three Dose Levels of AZD7594 by Assessment of Tmax of AZD7594
Description: Comparison of tmax (time to reach maximum plasma concentration) of AZD7594 on Day 1 of each treatment period; up to 6 samples were collected in each period (i.e. in participants with intensive pharmacokinetic assessments, at pre-dose and 15 and 30 minutes, and 1, 2, and 4 h post-dose)
Time Frame: as for outcome 16
Population: as for outcome 18
Measure: Median (Full Range); unit: Hour
Arm/Group | AZD7594 58 μg | AZD7594 250 μg | AZD7594 800 μg
Number analyzed (Participants) | 9 | 9 | 8
Hour | 0.25 [0.23 to 0.27] | 0.25 [0.25 to 0.50] | 0.25 [0.25 to 0.55]

22. Secondary Outcome: Rate and Extent of Absorption of Three Dose Levels of AZD7594 Following Multiple Dose Administration by Assessment of Tmax,ss of AZD7594
Description: Comparison of tmax,ss (time to reach maximum plasma concentration at steady state) of AZD7594 on Day 14 of each treatment period; up to 10 samples were collected in each period (i.e. in participants with intensive pharmacokinetic assessments, at pre-dose and 15 and 30 minutes, and 1, 2, 4, 8, 12, 16 and 24 h post-dose)
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Median (Full Range); unit: Hour
Arm/Group | AZD7594 58 μg | AZD7594 250 μg | AZD7594 800 μg
Number analyzed (Participants) | 9 | 9 | 8
Hour | 0.25 [0.25 to 0.50] | 0.25 [0.23 to 0.27] | 0.25 [0.25 to 0.98]

23. Secondary Outcome: Rate and Extent of Absorption of Three Dose Levels of AZD7594 Following Multiple Dose Administration by Assessment of Cavg,ss of AZD7594
Description: Comparison of Cavg,ss (average plasma concentration during a dosing interval at steady state) of AZD7594 on Day 14 of each treatment period; up to 10 samples were collected in each period (i.e. in participants with intensive pharmacokinetic assessments, at pre-dose and 15 and 30 minutes, and 1, 2, 4, 8, 12, 16 and 24 h post-dose)
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol/L
Arm/Group | AZD7594 58 μg | AZD7594 250 μg | AZD7594 800 μg
Number analyzed (Participants) | 9 | 9 | 8
pmol/L | 19.48 (17.93) | 71.89 (44.33) | 203.9 (52.55)

24. Secondary Outcome: Rate and Extent of Absorption of Three Dose Levels of AZD7594 Following Multiple Dose Administration by Assessment of Cmax/D of AZD7594
Description: Comparison of Cmax/D (dose-normalized Cmax) of AZD7594
Time Frame: On Day 1 in each period
Population: as for outcome 18
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol/L/μmol
Arm/Group | AZD7594 58 μg | AZD7594 250 μg | AZD7594 800 μg
Number analyzed (Participants) | 9 | 9 | 8
pmol/L/μmol | 380.8 (32.80) | 223.4 (34.17) | 128.5 (43.21)

25. Secondary Outcome: Rate and Extent of Absorption of Three Dose Levels of AZD7594 Following Multiple Dose Administration by Assessment of AUC(0-24)/D of AZD7594
Description: Comparison of AUC(0-24)/D (dose-normalized AUC(0-24)) of AZD7594
Time Frame: On Day 14 in each period
Population: as for outcome 18
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pmol/L/ μmol
Arm/Group | AZD7594 58 μg | AZD7594 250 μg | AZD7594 800 μg
Number analyzed (Participants) | 9 | 9 | 8
h*pmol/L/ μmol | 4886 (17.91) [3977 to 4944] | 4188 (44.33) | 3708 (52.48)

26. Secondary Outcome: Rate and Extent of Absorption of Three Dose Levels of AZD7594 Following Multiple Dose Administration by Assessment of Cmin of AZD7594
Description: Comparison of steady-state minimum (pre-dose) concentration (Cmin) of AZD7594 in each treatment period
Time Frame: On Day 14 at pre-dose in each period
Population: The subset of all randomized participants, 24-hour PK sampling was performed on Day 14, primary PK parameters (Cmax , AUC(0-4), Cmax,ss, AUC(0-24)) were calculated in at least one treatment period, and who had no major protocol deviations considered to impact the analysis of the PK data. Cmin was not determined for AZD7594 58 μg
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol/L
Arm/Group | AZD7594 58 μg | AZD7594 250 μg | AZD7594 800 μg
Number analyzed (Participants) | 9 | 9 | 8
pmol/L | NA (NA) — Not applicable for AZD7594 58 μg. Will be reported in the separate population PK report | 55.95 (51.74) | 191.6 (68.27)

ADVERSE EVENTS:
Time Frame: From Screening to Follow-up (these two examinations are up to 165 days apart)
Groups:
- Placebo (PBO): Placebo for AZD7594 DPI once daily
Arm/Group | Placebo (PBO) | AZD7594 58 μg | AZD7594 250 μg | AZD7594 800 μg
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/34 | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 17/52 | 13/34 | 9/34 | 12/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (PBO) (N=52) | AZD7594 58 μg (N=34) | AZD7594 250 μg (N=34) | AZD7594 800 μg (N=34)
Nasopharyngitis (Infections and infestations) | 8 | 4 | 2 | 4
Gastroenteritis (Infections and infestations) | 0 | 3 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 3 | 2
Migraine (Nervous system disorders) | 0 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 3
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0 | 1 | 0
Hepatosplenomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Anaemia vitamin B12 deficiency (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Eye irritation (Eye disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a publication (e.g., in a scientific journal) based on the results of this study is envisaged, approval from AstraZeneca will be obtained and a draft manuscript will be submitted to AstraZeneca for scrutiny and comment. The choice of conduit will be mutually agreed.